CLINICAL TRIAL: NCT00204841
Title: Rhinovirus Infection and Asthma in Childhood and Adolescents
Brief Title: Childhood Origins of Asthma (COAST)
Acronym: COAST
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1998-129; P01HL070831 (NIH); 2013-0144 (Other: UW IRB); H-2007-0044 (Other: UW IRB)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Asthma; Allergy
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasal mucus samples, cord blood, peripheral blood samples, nasal cell brushing samples, cell lines
Oversight: Data Monitoring Committee: No

SUMMARY:
Although asthma is likely to be a heterogeneous disease or syndrome, three factors and/or events repetitively emerge for their ability to significantly influence asthma inception in the first decade of life: immune response aberrations, which appear to be defined best by the concept of cytokine dysregulation; lower respiratory tract infections (in particular RSV); and some form of gene by environment interaction that needs to occur at a critical time period in the development of the immune system or the lung. It remains to be firmly established, however, how any one or all of these factors, either independently or interactively, influence the development of childhood asthma. Thus, our efforts to determine and define the importance of these three factors to asthma pathogenesis are the focus and goal of this current grant application.

DETAILED DESCRIPTION:
No more description necessary.

ELIGIBILITY:
Inclusion Criteria:

* children who had one or more parent with a history of allergy or asthma

Exclusion Criteria:

* pre term infants
* low birth weight infants
* respiratory distress at birth

Ages: 1 Minute to 2 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: High risk birth cohort of children (one or both parents have allergies and/or asthma).
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 1998-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the children longitudinally for the inception and progression of asthma. | Birth through age 19
  Clinical diagnosis of childhood asthma at age 6 years and older.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Jackson, MD, Principal Investigator — University of Wisconsin, Madison; Robert F Lemanske, Jr., MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- See also: study web page — http://www.medicine.wisc.edu/research/researchmain